CLINICAL TRIAL: NCT00720213
Title: Evaluation of Software Enhancements to the Respironics BiPAP autoSV Device
Brief Title: Evaluation of Software Enhancements to the Respironics BiPAP Auto Servo Ventilation (AutoSV) Device
Acronym: AUTOSV3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MR-0731-ASV3-MS
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Sleep Disordered Breathing; Sleep Apnea, Central
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respironics BiPAP autoSV2, Then Respironics BiPAP autoSV3 (Active Comparator): Participants will be randomized to receive Respironics BiPAP autoSV2 first and Respironics BiPAP autoSV3 second.
  Interventions: Device: Respironics BiPAP autoSV2; Device: Respironics BiPAP autoSV3
- Respironics BiPAP autoSV3, then Respironics BiPAP autoSV2 (Experimental): Participants will be randomized to receive Respironics BiPAP autoSV3 first and Respironics BiPAP autoSV2.
  Interventions: Device: Respironics BiPAP autoSV2; Device: Respironics BiPAP autoSV3

INTERVENTIONS:
Device: Respironics BiPAP autoSV2 — Respironics BiPAP autoSV2 is an Auto Servo Ventilation Device. This will be used on a randomized night.
Device: Respironics BiPAP autoSV3 — Respironics BiPAP autoSV3 is an Auto Servo Ventilation Device. This will be used on a randomized night.
  Other Names: Respironics BiPAP autoSV3 advanced

SUMMARY:
This study is being undertaken to collect data from Respironics Inc's BiPAP Auto Servo Ventilation 3 (autoSV3) and compare with data from Respironics, Inc's BiPAP autoSV2, to confirm that the algorithms in the BiPAP autoSV3 device can safely and effectively treat participants experiencing Complex Sleep Apneas (Comp SAS) no worse than its predecessor, the BiPAP auto Servo ventilation 2 (autoSV2) device. This will be determined using a comparative, randomized design with the participants blinded to the therapy. Additionally, attempts will be made to blind the central scorer(s) with respect to which device is in use.

DETAILED DESCRIPTION:
This study was conducted to evaluate the therapeutic performance of a new auto Servo Ventilation device (Philips Respironics autoSV Advanced) for the treatment of complex central sleep apnea (CompSA). The features of autoSV Advanced include an automatic expiratory pressure (EPAP) adjustment, an advanced algorithm for distinguishing open versus obstructed airway apnea, a modified auto backup rate which is proportional to subject's baseline breathing rate, and a variable inspiratory support. Our primary aim was to compare the performance of the advanced servo-ventilator (BiPAP autoSV Advanced) with conventional servo-ventilator (BiPAP autoSV) in treating central sleep apnea (CSA).

Study Design: A prospective, multicenter, randomized, controlled trial.

Setting: Five sleep laboratories in the United States.

Participants: Thirty-seven participants were included.

ELIGIBILITY:
Inclusion Criteria:

Pre-Study Inclusion Criteria:

* Age 21-80
* Ability to provide consent
* Documentation of medical stability by investigator

Enrollment Inclusion Criteria:

• Participants who, during the ambulatory polysomnography (PSG) study (Stardust), or in lab Diagnostic PSG demonstrated an Apnea Hypopnea Index (AHI) ≥10 or Central Apnea Index (CAI) ≥5

or

• Participants who previously demonstrated Central sleep Apnea (CSA), with a CAI≥5 on Continuous Positive Airway Pressure (CPAP) titration.

Exclusion Criteria:

* • Participants who are acutely ill, medically complicated or who are medically unstable.

  * Pregnancy (will confirm absence of pregnancy with a urine or serum pregnancy test in women of child bearing potential).
  * Participants in whom PAP therapy is otherwise medically contraindicated.
  * Participants who are unwilling to wear CPAP
  * Participants who are currently prescribed nocturnal oxygen use and are unable to forego oxygen during study nights.
  * Participants with previously diagnosed respiratory failure or respiratory insufficiency and who are known to have chronically elevated arterial carbon dioxide levels while awake (PaCO2 ≥ 45mmHg).
  * Participants who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
  * Participants with untreated, non- Obstructive Sleep Apnea (OSA)/CSA sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome (PLM Arousal Index > 15).
  * Participants who are unwilling to participate in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Goodwin, Principal Investigator — University of Arizona; Shahrokh Javaheri, MD, Principal Investigator — Sleepcare Diagnostics; Rami Khayat, MD, Principal Investigator — Ohio State Univercity; Mark Goetting, MD, Principal Investigator — Sleep Health; Paul Wylie, MD, Principal Investigator — Arkansas Center for Sleep Medicine
Locations (5):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - Mark G. Goetting, Portage, Michigan
  - Ohio State University, Columbus, Ohio
  - Sleepcare Diagnostics, Mason, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the investigators' sleep labs.
Pre-assignment Details: Participants were excluded if they did not demonstrate an Apnea-Hypopnea Index (AHI) ≥ 10 and Central Apnea Index (CAI)≥ 5 during the diagnostic polysomnography (PSG), or if they did not demonstrate a CAI ≥ 5 on continuous positive airway pressure (CPAP) titration.
Groups:
- Screening Phase: All participants that signed a consent form.
- BiPap Auto SV2 Device First, BiPap Auto SV3 Device Second: BiPAP auto servo ventilation (SV) 2 Device. This arm used the BiPAP AutoSV2 overnight first overnight, followed by the BiPAP auto servo ventilation (SV) 3 Device. This arm used the BiPAP AutoSV3 for the second overnight.
- BiPap Auto SV3 Device First, BiPap AutoSV2 Device Second: BiPAP auto servo ventilation (SV) 3 Device. This arm used the BiPAP AutoSV3 for the first overnight. The second overnight participants used the BiPap Auto Servo Ventilation 2 Device.
Period: Screening Phase With Diagnostic PSG
Arm/Group | Screening Phase | BiPap Auto SV2 Device First, BiPap Auto SV3 Device Second | BiPap Auto SV3 Device First, BiPap AutoSV2 Device Second
Started | 44 | 0 | 0
Completed | 37 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Screen Failure | 7 | 0 | 0
Period: Treatment Period
Arm/Group | Screening Phase | BiPap Auto SV2 Device First, BiPap Auto SV3 Device Second | BiPap Auto SV3 Device First, BiPap AutoSV2 Device Second
Started | 0 | 20 | 17
Completed | 0 | 20 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who met inclusion/exclusion criteria were included in the baseline analysis.
Groups:
- All Study Participants: Participants who signed the informed consent
Arm/Group | All Study Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 37
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31 (6)

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index
Description: The number of apneas and hypopneas per hour of sleep. Apneas are the cessation of airflow at the nostrils and mouth for at least 10 seconds as determined using nasal-oral thermistor or device flow. Hypopneas is shallow breathing in which the air flow in and out of the airway is significantly reduced as detected by nasal pressure or device flow - often associated with oxygen desaturation of 4% or EEG arousal.
  A central sleep scorer was utilized to review of the overnight PSGs and count the number of apneas and hyopneas per hour. The index is the average number for apneas+hyopneas per hour.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Respironics BiPAP autoSV2: Respironics BiPAP autoSV2
- Respironics BiPAP autoSV3: Respironics BiPAP autoSV3
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events/hour | 10.44 (10.3) | 6.06 (5.81)
Statistical Analysis 1: Comparison: Respironics BiPAP autoSV2 vs Respironics BiPAP autoSV3; Each participant was treated with the BiPAP autoSV2 (ASV2) and autoSV Advanced (ASV3) on two separate nights; therefore, the data were analyzed as paired samples. Depending on normality, each endpoint was analyzed with either a paired t-test or the nonparametric Wilcoxon Signed Ranks test. All comparisons were 2-sided conducted at a 5% level of significance; Test type: Superiority or Other; p = 0.0054, Wilcoxon Signed Rank test; Mean Difference (Final Values) = 3.98, 95% CI 2-sided [1.44 to 6.51], Standard Deviation 8.03

2. Secondary Outcome: Apnea Hypopnea Index- REM and NREM
Description: The number of apneas and hypopneas per hour of sleep while in REM (rapid eye movement) and in NREM (non-rapid eye movement)
  A central sleep scorer was utilized to review of the overnight PSGs and count the number of apneas and hyopneas per hour while in REM vs. NREM.
Time Frame: 2 nights
Population: Data was not scorable for NREM.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events/hour
  Apnea Hypopnea Index- REM: number analyzed (Participants) | 36 | 35
  Apnea Hypopnea Index- REM | 3.27 (6.15) | 2.09 (3.74)
  Apnea Hypopnea Index- NREM | 6.84 (6.52) | 11.74 (11.70)

3. Secondary Outcome: Central Apnea Index
Description: The number of central apneas divided by the number of hours of sleep. Central apneas are the cessation of airflow at the nostrils and mouth for at least 10 seconds that is associated with the absence of inspiratory effort.
  A central sleep scorer was utilized to review of the overnight PSGs and count the number of central apneas per hour.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events/hour | 2.82 (3.72) | 0.56 (.71)

4. Secondary Outcome: Obstructive Apnea Index
Description: Obstructive sleep apnea (OSA) is the most common type of sleep apnea and is caused by complete or partial obstructions of the upper airway.
  A central sleep scorer was utilized to review of the overnight PSGs and count the number of obstructive apneas per hour.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events/hour | 2.04 (2.35) | 1.14 (1.59)

5. Secondary Outcome: Mixed Apnea Index
Description: Mixed sleep apnea is a combination of both obstructive and central sleep apnea symptoms
  A central sleep scorer was utilized to review of the overnight PSGs and count the number of mixed apneas per hour.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events/hour | 0.44 (.69) | 0.20 (0.37)

6. Secondary Outcome: Hypopnea Index
Description: Hypopneas are characterized by shallow breathing in which the air flow in and out of the airway is significantly reduced as detected by nasal pressure or device flow - often associated with oxygen desaturation of 4% or EEG arousal.
  A central sleep scorer was utilized to review of the overnight PSGs and count the number of hyopneas per hour.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events/hour | 5.11 (6.22) | 4.16 (4.97)

7. Secondary Outcome: Sleep Onset Latency
Description: Sleep onset latency is the length of time that it takes to accomplish the transition from full wakefulness to sleep, normally to the lightest of the non-REM sleep stages. This found by reviewing the number of minutes in the PSG it took from lights off until the lightest non-REM sleep.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
minutes | 18.91 (18.53) | 20.91 (16.76)

8. Secondary Outcome: Rapid Eye Movement (REM) Onset Latency
Description: Rapid eye movement latency is the time from the sleep onset to the first epoch of REM sleep; therefore, it depends on the patient's sleep latency.
Time Frame: 2 nights
Population: This data was not part of the scoring PSG criteria and therefore not collected.
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Wake After Sleep Onset
Description: Wake after sleep onset refers to periods of wakefulness occurring after defined sleep onset. This was calculated by adding the total number of minutes the participant was awake after sleep onset.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
minutes | 88.67 (52.33) | 93.47 (58)

10. Secondary Outcome: Total Sleep Time
Description: Total sleep time is the total time the participant was asleep after sleep onset. This is calculated by adding the total number of minutes the participant was asleep during the night after sleep onset.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
minutes | 361.23 (72.55) | 370.59 (61.19)

11. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency is a measure of how much a participant slept over the night. This is calculated by comparing the total sleep time and the total recording time * 100.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: percentage efficiency
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
percentage efficiency | 76.84 (13.39) | 76.46 (11.93)

12. Secondary Outcome: Stages N1,N2,N3 (NREM), and REM (R) Sleep (in Minutes)REM, NREM and Total Sleep Time.
Description: These measures are the amount of time patients spent in each stage of sleep in minutes.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
minutes
  Stage 1 | 16.72 (11.79) | 16.02 (9.19)
  Stage 2 | 54.54 (11.62) | 55.06 (11.99)
  Stage 3 | 13.25 (9.81) | 11.75 (10.29)
  REM | 15.5 (6.35) | 17.18 (7.43)
  TST | 361.23 (72.55) | 370.59 (61.19)

13. Secondary Outcome: Wake (W), Stages N1,N2,N3 (NREM), and REM (R) Sleep (% TST)
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
minutes
  Stage 1 | 16.72 (11.79) | 16.02 (9.19)
  Stage 2 | 54.54 (11.62) | 55.06 (11.99)
  Stage 3 & 4 | 13.25 (9.81) | 11.75 (10.29)
  REM | 15.50 (6.35) | 17.18 (7.43)

14. Secondary Outcome: Arousal Index [Total, Apnea Hypopnea (AH)-Related, Periodic Limb Movement (PLM)-Related, 'Spontaneous']
Description: The number of arousals and awakenings is registered in the study, and reported as a total number and as a frequency per hour of sleep, which is referred to as an index. The higher the arousal index, the more tired you are likely to feel, though people vary in their tolerance of sleep disruptions.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 37 | 37
events per hour | 26.04 (11.11) | 23.58 (10.59)

15. Secondary Outcome: Nocturnal Oxygenation (Measured by Continuous Pulse Oximetry During Sleep Study)
Description: Measure of oxygen saturation as measured by a pulse oximetry over the course of the night.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Treatment Group 1: Respironics BiPAP autoSV2
- Treatment Group 2: Respironics BiPAP autoSV3
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 37 | 37
percentage of oxygen saturation
  Baseline Nocturnal oxygenation (%) | 95.78 (1.18) | 95.7 (1.43)
  Lowest Nocturnal oxygenation (%) | 86.54 (8.74) | 87.84 (4.60)

16. Secondary Outcome: Apnea Hypopnea Index (REM, NREM and TST) Using Modified Hypopnea Rule.
Description: This is the measure of the Apnea Hypopnea Index as measured by using a modified hypopnea rule. The modified hypopnea rule is a scoring change when AHI changes due to central vs obstructive apneas.
Time Frame: 2 nights
Population: During scoring of the PSG the modified hypopnea rule wasn't utlized therefore this data is not provided.
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Apnea Hypopnea Index(REM, NREM and TST) During Epochs for Which Leak is Determined to Exist Within Acceptable Limits.
Description: The AHI during epochs for which leak is determined to exist within acceptable limits occurs is the same calculation during AHI is normally calculated just in a 30 second (epoch) time period.
Time Frame: 2 nights
Population: This was not part of the standard scoring of the PSG, therefore this was not calculated
Arm/Group | Respironics BiPAP autoSV2 | Respironics BiPAP autoSV3
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Treatment Group 1: BiPAP autoSV2 Device
- Treatment Group 2: BiPAP autoSV3 Device
Arm/Group | Treatment Group 1 | Treatment Group 2
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
Not all of the secondary analysis was completed as this study also captured engineering data which is not part of standard PSG scoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days